CLINICAL TRIAL: NCT03490240
Title: Project BIPAMS: Behavioral Intervention for Physical Activity in Multiple Sclerosis
Acronym: BIPAMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Donald Lein, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 170609001
Record Dates: First submitted 2018-01-23; First posted 2018-04-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The investigators will advertise the study as comparing two approaches delivered through the Internet for managing consequences of MS and improving health indicators. On randomization, the investigators will again reaffirm this position with the participant. The participant will not be informed about which condition is the control or the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIPAMS (Experimental): The behavioral intervention consists of two primary components, a dedicated Internet website and one-on-one video chats with a behavioral coach via Skype. The behavioral intervention focuses on the skills, techniques, resources, and strategies for becoming and staying physically active with MS, but it does not provide a prescription for exercise or physical activity itself.
  Interventions: Behavioral: BIPAMS
- WELLMS (Active Comparator): The control condition provides an Internet website and one-on-one video chats that discuss materials about self-managing MS consequences and health indicators through methods other than physical activity.
  Interventions: Behavioral: WELLMS

INTERVENTIONS:
Behavioral: BIPAMS — The primary content of the website is delivered through interactive video courses. The interactive video courses are released seven times during the first two months, four times during the second two months, and twice during the final two months of the intervention.
  Another key part of the website is the Tracker feature. This feature allows for tracking of daily step counts (via Yamax SW-200 pedometer) as well as setting goals and monitoring progress over the program.
  The one-on-one video chats are conducted face to face through skype and are semi-scripted. The chats consist of an ongoing review of goal-setting and progress toward goal attainment through Tracker as well as discussion of strategies and facilitators of behavioral change based on SCT and current website content. The chats occur seven times during the first two months, four times during the second two months, and twice during the final two months of the intervention.
  Arms: BIPAMS
Behavioral: WELLMS — The control condition focuses on self-managing MS through means other than physical activity. The materials are transformations of brochures provided by the NMSS, including Gait or Walking Problems: The Basic Facts; MS and Your Emotions; Pain: The Basic Facts; Solving Cognitive Problems; Taming Stress in MS; Food for Thought: MS and Nutrition; and Vitamins, Minerals, and Herbs: An Introduction. The delivery of the Internet materials and chat sessions will occur on the same time schedule and frequency as the intervention condition, and will have a comparable time commitment. The control condition will account for attention and social contact as well as other possible biases such as initial reactivity and time spent on the website and video chats. The participants in the control condition will not be offered the behavioral intervention for increasing physical activity after completion of the study procedures.
  Arms: WELLMS

SUMMARY:
This randomized controlled trial will examine the effect of a 6-month behavioral intervention, based on social cognitive theory and delivered through the Internet, for increasing physical activity and secondarily improving mobility, cognition, symptoms and quality of life in persons with MS. The investigators hypothesize that individuals who receive the 6-month behavioral intervention will demonstrate an increase in physical activity behavior that will last throughout a 6-month follow up compared with participants in the control condition. The investigators further hypothesize that individuals in the behavioral intervention will demonstrate better walking mobility and cognitive function, reduced fatigue, depression, anxiety, and pain, and improved quality of life compared to the control condition. The investigators hypothesize that the behavioral intervention will increase physical activity through positive changes in self-efficacy, outcome expectations, goal setting, and impediments as social-cognitive determinants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* Relapse free in the past 30 days
* Internet and email access
* Willingness to complete the questionnaires, wear the accelerometer, and undergo randomization
* Being non-active defined as not engaging in regular activity (30 minutes accumulated per day) on more than 2 days of the week during the previous six months
* Ability to ambulate with or without assistance (i.e. walking with or without a can or walker, but not a wheelchair)
* Age between 18 and 64

Exclusion Criteria:

* Moderate or high risk for undertaking strenuous or maximal exercise per participants response to the PAR-Q. Those who report no more than one YES or affirmative on the 7 item PAR-Q will be considered at low risk and included for participation. All others will be considered at moderate or high risk and excluded from participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Physical Activity levels through Accelerometery from baseline at 6 and 12 months. | Baseline through 12 months
  Physical activity will be assessed using an ActiGraph accelerometer. Participants will wear an accelerometer on a belt around their waist during the waking hours of a 7 day period. Participants will complete this at baseline, 6 months, and 12 months.
Change of Physical Activity levels through the Godin Leisure-Time Exercise Questionnaire from baseline at 6 and 12 months. | Baseline through 12 months.
  Physical activity will be assessed using the Godin Leisure-Time Exercise Questionnaire. Participants will complete this questionnaire at baseline, 6 months, and 12 months.
Change of Physical Activity levels through the Abbreviated International Physical Activity Questionnaire from baseline at 6 and 12 months. | Baseline through 12 months.
  Physical activity will be assessed using the Abbreviated International Physical Activity Questionnaire. Participants will complete this questionnaire at baseline, 6 months, and 12 months.

SECONDARY OUTCOMES:
Change of self-report measures of walking through the Multiple Sclerosis Walking Scale - 12 from baseline at 6 and 12 months | Baseline through 12 months
  Self report measures of walking will be assessed through the Multiple Sclerosis Walking Scale - 12. Participants will complete this questionnaire at baseline, 6 month, and 12 months.
Change of self-report measures of Walking through the Patient Determined Disease Steps Scale from baseline at 6 and 12 months. | Baseline through 12 months
  Self report measures of walking will be assessed through the Patient Determined Disease Steps Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months.
Change of self-report measures of Cognition through the Perceived Deficits Questionnaire from baseline at 6 and 12 months. | Baseline through 12 months
  Self report measures of cognition will be assessed through the Perceived Deficits Questionnaire. Participants will complete this questionnaire at baseline, 6 month, and 12 months.
Change of self-report measures of Cognition through the Multiple Sclerosis Neuropsychological Questionnaire from baseline at 6 and 12 months. | Baseline through 12 months
  Self report measures of cognition will be assessed through the Multiple Sclerosis Neuropsychological Questionnaire. Participants will complete this questionnaire at baseline, 6 month, and 12 months.
Change of self-report measures of Fatigue through the Fatigue Severity Scale from baseline at 6 and 12 months. | Baseline through 12 months
  Self report measures of fatigue will be assessed through the Fatigue Severity Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Change of self-report measures of Fatigue through the Modified Fatigue Impact Scale at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures of fatigue will be assessed through the Modified Fatigue Impact Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Change of self-report measures of Anxiety and Depression through the Hospital Anxiety and Depression Scale at 6 months and 12 months from baseline. | Baseline through 12 months
  Self report measures of Anxiety and Depression will be assessed through the Hospital Anxiety and Depression scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Change of self-report measures of Pain through the Short-form of McGill Pain Questionnaire at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures of Pain will be assessed through the Short-form of McGill Pain Questionnaire. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures of sleep through the Pittsburgh Sleep Quality Index at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures of sleep will be assessed through the Pittsburgh Sleep Quality Index. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures of quality of life through the Medical Outcomes Study Short Form-36 at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures of quality of life will be assessed through the Medical Outcomes Study Short Form-36 . Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures of quality of life through the Multiple Sclerosis Impact Scale-29 at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures of quality of life will be assessed through the Multiple Sclerosis Impact Scale-29. Participants will complete this questionnaire at baseline, 6 month, and 12 months

OTHER OUTCOMES:
Changes of self-report measures based on Social Cognitive Theory on Self-Efficacy through the MS Self-Efficacy Sale at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for self-efficacy will be assessed through the MS Self-Efficacy scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures based on Social Cognitive Theory on Self-Efficacy through the Exercise Self-Efficacy Scale at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for self-efficacy will be assessed through the Exercise Self-Efficacy Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures based on goal setting through the Exercise Goal Setting and Planning Scale at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for goal setting will be assessed through the Exercise Goal Setting and Planning Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures based on outcome expectations through the Multidimensional Outcome Expectancies for Exercise Scale at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for outcome expectations will be assessed through the Multidimensional Outcome Expectancies for Exercise Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures based on quality of life through the Late-Life Function and Disability Inventory at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for quality of life will be assessed through the Late-Life Function and Disability Inventory. Participants will complete this questionnaire at baseline, 6 month, and 12 months
Changes of self-report measures based on quality of life through the Social Provisions Scale Inventory at 6 and 12 months from baseline. | Baseline through 12 months
  Self report measures for quality of life will be assessed through the Social Provisions Scale. Participants will complete this questionnaire at baseline, 6 month, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lein, PhD, Principal Investigator — Associate Professor
Locations (1):
- Exercise Neuroscience Research Lab, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Motl RW, Kidwell-Chandler A, Sandroff BM, Pilutti LA, Cutter GR, Aldunate R, Bollaert RE. Primary results of a phase-III, randomized controlled trial of the Behavioral Intervention for increasing Physical Activity in Multiple Sclerosis project. Mult Scler. 2023 Mar;29(3):415-426. doi: 10.1177/13524585221146430. PMID 36843446
- [Derived] Motl RW, Sandroff BM, Pilutti LA, Cutter GR, Aldunate R, Kidwell-Chandler A, Bollaert RE. Randomized controlled trial of the behavioral intervention for increasing physical activity in multiple sclerosis project: Secondary, patient-reported outcomes. Contemp Clin Trials. 2023 Feb;125:107056. doi: 10.1016/j.cct.2022.107056. Epub 2022 Dec 16. PMID 36535606
- [Derived] Silveira SL, McCroskey J, Wingo BC, Motl RW. eHealth-Based Behavioral Intervention for Increasing Physical Activity in Persons With Multiple Sclerosis: Fidelity Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Mar 1;8(3):e12319. doi: 10.2196/12319. PMID 30821692